CLINICAL TRIAL: NCT03770676
Title: Investigating Flavour-nutrient Learning in Humans Using Novel-flavoured, Selenium-fortified Biscuits
Brief Title: Investigating the Sensory Attributes of Selenium-fortified Biscuits and Their Effects on Selenium-status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Fera Science Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1533/4994/2018
Record Dates: First submitted 2018-09-20; First posted 2018-12-10 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-10

CONDITIONS: Selenium Status
Keywords: Food sensory perception; Selenium

STUDY DESIGN:
Intervention Model Description: There are three study groups (three 'test' biscuit flavours). Each study group will be assigned one test flavour ('intervention' flavour/biscuit). They begin consumption of their intervention biscuits on day 1 and finish on day 14. Plasma selenium concentration and sensory perception of biscuits will be measured on day 1 (baseline), 8 (post-7 days of intervention) and 15 (post-14 days of intervention).
Who Masked: Participant, Investigator
Masking Description: The investigator will be blinded to which (intervention) flavour each participant is assigned to.
  Both the investigator and the participant will be blinded to the participant's plasma selenium concentration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flavour 1 (Experimental): Selenium-fortified biscuits These participants will be assigned to biscuit flavour 1. If possible, there will be an equal number of low, medium and high selenium-status participants. They will consume this flavour of selenium-fortified biscuits for 14 consecutive days at home, providing approximately 60 mcg selenium per day.
  Interventions: Dietary Supplement: Selenium-fortified biscuits
- Flavour 2 (Experimental): Selenium-fortified biscuits These participants will be assigned to biscuit flavour 2. If possible, there will be an equal number of low, medium and high selenium-status participants. They will consume this flavour of selenium-fortified biscuits biscuit for 14 consecutive days at home, providing approximately 60 mcg selenium per day.
  Interventions: Dietary Supplement: Selenium-fortified biscuits
- Flavour 3 (Experimental): Selenium-fortified biscuits These participants will be assigned to biscuit flavour 3. If possible, there will be an equal number of low, medium and high selenium-status participants. They will consume this flavour of selenium-fortified biscuits for 14 consecutive days at home, providing approximately 60 mcg selenium per day.
  Interventions: Dietary Supplement: Selenium-fortified biscuits

INTERVENTIONS:
Dietary Supplement: Selenium-fortified biscuits — Selenium-fortified biscuits, fortified with selenium-enriched yeast (approx. 60 mcg selenium per day, for 14 days). One of three novel flavours.

SUMMARY:
This intervention study will investigate the relationship between consumption of selenium-fortified biscuits fortified with selenium-enriched yeast (approximately 60mcg of selenium per day for 14 days) and both plasma selenium concentration and plasma selenoprotein P concentration in adult human volunteers. It will also investigate how selenium-status may affect changes in sensory perception of the fortified biscuits when consumed for 7 and 14 consecutive days (Flavour-Nutrient Learning).

DETAILED DESCRIPTION:
There are different forms of selenium supplementation which may be used to improve selenium-status, one being selenium-enriched yeast.

Selenium is an essential micronutrient consumed through food, however the selenium contents of foods is variable, and depends upon the soil the food has been grown in. The UK population may not consume enough selenium through their diet, due to selenium levels in British soil being low and the use of North American wheat flour being increasingly replaced with lower selenium European flour.

It is therefore relevant to explore the ability of selenium-enriched yeast to improve selenium status if initially low. It is also important to investigate if the sensory attributes of selenium-fortified foods are different to unfortified foods. Additionally, investigating Flavour-Nutrient Learning (how selenium-status might change sensory perception of selenium-rich foods) could improve understanding of food choices.

This study aims to investigate the following topics:

1. The relationship between selenium intake (through selenium-fortified biscuits) and selenium-status.
2. How selenium-status affects sensory perception of selenium-fortified biscuits (Flavour Nutrient Learning, FNL).

ELIGIBILITY:
Inclusion Criteria:

1. Adult human volunteers, 18 years of age or older.
2. Generally healthy, meaning that if health issues such as hypertension, diabetes, arthritis etc. are present, they are well controlled by appropriate treatments.
3. Upon tasting the screening biscuit, are confident they would be able to eat the specified amount every day for 14 consecutive days.
4. No taste or smell disorders.
5. No difficulties with chewing and/or swallowing.
6. No intolerances and/or allergies to any of the test foods.
7. No impairments which may prevent mental understanding of the trial, or informed consent from being given.
8. No disorders/medication that would make blood sampling dangerous to their health.
9. Plasma selenium not lower than 28 µg/L or higher than 400 µg/L on analysis
10. Participants need to be able to visit Newcastle University for the scheduled visits.
11. Participants must have been living in the UK for at least 6 months.

Exclusion Criteria:

Do not meet all requirements in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in preference for the intervention flavour over two other test flavours and plain flavour, after 14 days of consumption of Se-fortified intervention-flavoured biscuits. | Day 1 (baseline) and day 15 (post-14 days of intervention biscuit consumption).
  Participants score their intervention flavour (the test flavour they eat for 14 days), two test flavours (not eaten for 14 days) and plain flavour using a visual analogue scale anchored by "not very"/0 and "very"/100. They do this for liking of smell, taste, texture, aftertaste and pleasantness of the overall eating experience. This is repeated three times (three plates of biscuits) in one food sensory test. Each attribute for each plate will have a 'preference score' calculated, using the following equation:
  Preference score = (score of intervention flavour) - (average score of other 3 flavours).
  Preference scores are then averaged across the three plates.
  Flavour preference change is calculated as the change in average flavour preference score from baseline (day 1 food sensory test) to after 14 days of intervention biscuit consumption at home (day 15 food sensory test):
  Preference change = day 15 score - day 1 score

SECONDARY OUTCOMES:
Change in preference for the intervention flavour over two other test flavours and plain flavour, after 7 days of consumption of Se-fortified biscuits flavoured with the intervention flavour. | Day 1 (baseline) and day 8 (post 7 days of intervention biscuit consumption).
  Preference scores for each day are calculated using the formula in the primary outcome measure. Preference change is calculated using the following formula:
  Preference change = day 8 score - day 1 score
Change in preference for the intervention flavour over two other test flavours, after 14 days of consumption of Se-fortified biscuits flavoured with the intervention flavour. | Day 1 (baseline) and day 15 (post 14 days of intervention biscuit consumption).
  Preference scores for each day are calculated using the formula in the primary outcome measure, except without including the scores of the plain flavour. Preference change is measured using the formula in the primary outcome measure.
Change in preference for the intervention flavour over two other test flavours, after 7 days of consumption of Se-fortified biscuits flavoured with the intervention flavour. | Day 1 (baseline) and day 8 (post 7 days of intervention biscuit consumption).
  Preference scores for each day are calculated using the formula in the primary outcome measure, except without including the scores of the plain flavour. Preference change is measured using the formula in the second outcome measure.
Change in preference for the intervention flavour over plain flavour, after 14 days of consumption of Se-fortified biscuits flavoured with the intervention flavour. | Day 1 (baseline) and day 15 (post 14 days of intervention biscuit consumption).
  Preference scores for each day are calculated using the formula in the primary outcome measure, except without including the scores of the two test flavour. Preference change is measured using the formula in the primary outcome measure.
Change in preference for the intervention flavour compared with plain flavour, after 7 days of consumption of Se-fortified biscuits flavoured with the intervention flavour. | Day 1 (baseline) and day 8 (post 7 days of intervention biscuit consumption).
  Preference scores for each day are calculated using the formula in the primary outcome measure, except without including the scores of the two test flavours. Preference change is measured using the formula in the second outcome measure.
Change in plasma selenium concentration after consumption of selenium-fortified biscuits (approximately 60 micrograms of selenium per day) daily for 14 consecutive days. | Day 1 (baseline) and day 15 (post 14 days of intervention biscuit consumption).
  Blood samples taken via venepuncture or finger-prick, centrifuged and plasma collected. Plasma analysed using inductively coupled plasma mass spectrometry (ICP-MS) after acid digestion.
  Change in plasma selenium concentration = concentration at day 15 (post 14 days of intervention biscuit consumption) - concentration at day 1 (baseline).
Change in plasma selenium concentration after consumption of selenium-fortified biscuits (approximately 60 micrograms of selenium per day) daily for 7 consecutive days. | Day 1 (baseline) and day 8 (post 7 days of intervention biscuit consumption).
  Blood samples taken via venepuncture or finger-prick, centrifuged and plasma collected. Plasma analysed using ICP-MS after acid digestion.
  Change in plasma selenium concentration = concentration at day 8 (post 7 days of intervention biscuit consumption) - concentration at day 1 (baseline).
Change in plasma selenoprotein P (SEPP1) concentration after consumption of selenium-fortified biscuits (approximately 60 micrograms of selenium per day) daily for 14 consecutive days. | Day 1 (baseline) and day 15 (post 14 days of intervention biscuit consumption).
  Blood samples taken via venepuncture, centrifuged and plasma collected. Plasma analysed using ELISA.
  Change in plasma selenoprotein P concentration = concentration at day 15 (post 14 days of intervention biscuit consumption) - concentration at day 1 (baseline).
Change in plasma selenoprotein P (SEPP1) concentration after consumption of selenium-fortified biscuits (approximately 60 micrograms of selenium per day) daily for 7 consecutive days. | Day 1 (baseline) and day 8 (post 7 days of intervention biscuit consumption).
  Blood samples taken via venepuncture, centrifuged and plasma collected. Plasma analysed using ELISA.
  Change in plasma selenoprotein P concentration = concentration at day 8 (post 7 days of intervention biscuit consumption) - concentration at day 1 (baseline).
How many participants prefer a fortified test biscuit over an unfortified version of their intervention biscuit in a paired comparison test? | Day 1 (baseline), day 8 (post-7 days intervention) and day 15 (post-14 days intervention).
  Participants are asked to indicate which they prefer from two biscuits on a plate. One biscuit will be a selenium-fortified test biscuit, and the other an unfortified version of their intervention biscuit. This is to test if preference is stronger for the intervention flavour or the Se-enriched yeast.
How many participants prefer a fortified test biscuit over an unfortified test biscuit of a different flavour in a paired comparison test? | Day 1 (baseline), day 8 (post-7 days intervention) and day 15 (post-14 days intervention).
  Participants are asked to indicate which they prefer from two biscuits on a plate. The biscuits will be the participant's two test flavours, one of which will be fortified. This is to test if a preference has developed for Se-enriched yeast flavour.
How many participants prefer their fortified intervention biscuit over an unfortified test biscuit in a paired comparison test? | Day 1 (baseline), day 8 (post-7 days intervention) and day 15 (post-14 days intervention).
  Participants are asked to indicate which they prefer from two biscuits on a plate. The biscuits will be the participant's fortified intervention biscuit, and an unfortified test biscuits. This is to test if participants prefer their intervention biscuit.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Brandt, PhD, Principal Investigator — Newcastle University
Locations (1):
- NU-Food, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided